CLINICAL TRIAL: NCT05359757
Title: Effect of Naturalistic Teaching Strategies in Children With Autism Spectrum Disorder
Brief Title: Naturalistic Teaching Strategies in Children With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/Lhr/21/0627 Maha Nasir
Record Dates: First submitted 2022-01-08; First posted 2022-05-04 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Naturalistic therapeutic techniques and PECS therapy. (Experimental)
  Interventions: Other: Effect of Naturalistic Teaching Strategies in Children with autism spectrum disorder; Other: PECS Therapy only
- PECS therapy Only. (Active Comparator)
  Interventions: Other: PECS Therapy only

INTERVENTIONS:
Other: Effect of Naturalistic Teaching Strategies in Children with autism spectrum disorder — In this group, the patients will be provided with both the naturalistic therapeutic techniques the PECS Therapy.
  A baseline of the kids in this group will be made using the portage guide and PECS
  * Incidental teaching trial, natural language paradigm, and time delay concepts will be incorporated in the therapy sessions and communication using picture cards will be made.
  * 40 minutes session will be conducted in which 20 minutes session will be for naturalistic teaching techniques and 20 minutes will be for PECS.
  * This will be followed for 30 sessions
  Arms: Naturalistic therapeutic techniques and PECS therapy.
Other: PECS Therapy only — A baseline will be developed using the portage guide and PECS.
  * Communication strategies using the PECS picture cards will be made
  * 30 minutes session will be conducted
  * This will be followed for 30 sessions

SUMMARY:
The study will show the effect of naturalistic teaching strategies and picture exchange communication systems in children with an autism spectrum disorder. There will be two groups in this study. One control group and the other experimental group.

One group will be provided with the naturalistic teaching strategies and pecs therapy both and the other group will be provided with the PECS therapy. The research will be conducted within the duration of six months after the approval from BASR.

The two groups will be first assessed using the portage early education program and pecs manual. After 20 sessions of respective therapeutic techniques, both of the groups will be reassessed. The results of both of the groups will be then compared and conclusions will be drawn.

DETAILED DESCRIPTION:
The Naturalistic Teaching approach is both adaptive and reactive to the needs of the kids with autism. Its methods are designed to be incorporated into the routines of children with an autism spectrum disorder. The naturalistic methods are intended to mimic the natural instructions a child receives in a variety of contexts.

PictureExchange Communication System (PECS) is a unique communication training program that was developed as a means of evading some shortcomings associated with these strategies. Many individuals with autism are candidates for augmentative and alternative communication (AAC) systems, either to supplement (i.e., augment) their existing speech or to act as their primary (i.e., alternative) method of expressive communication. Presently, aided, picture-based AAC systems are used more frequently and successfully with individuals with ASD. PECS consists of six phases and begins by teaching an individual to give a single picture of a desired item or action to a "communicative partner" who immediately honors the exchange as a request.

ELIGIBILITY:
Inclusion Criteria:

* Children who will be diagnosed with autism spectrum disorder and with speech and language impairments and will fall in the chronological age of language development (3-8) years
* Both genders
* Children who will have a vocabulary of 0-10 meaningful words
* Children with mild and moderate autism

Exclusion Criteria:

Children already taking speech therapy sessions

* Children with severe to a profound level.
* Children with any other disorder along with autism

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2021-11-25 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-04-10 (Actual)

PRIMARY OUTCOMES:
Portage Early Education Program for Naturalistic Teaching Strategies for children with autism spectrum disorder. | 30 Sessions (2 Months)
  Portage Guide to Early Education is a naturalistic teaching strategy. It consists of a set of reading materials and a method of training parents to teach their own children.It is a valid and reliable tool and is used in clinics as an assessment method. These strategies are treatment procedures in the natural environment, and promotes motivation, functional relationships, generalization and maintenance for children with autism spectrum disorder. The four parts of this technique includes: Natural Language Paradigm, Speech/Play Enhancement for Autistic Kids, Multiple Incidental Teaching Sessions, and Time Delay. These training procedures are incorporate components and strategies which are known to facilitate acquisition, generalization and maintenance of new behaviors. This teaching strategies are designed for therapists, parents and siblings.
Picture Exchange Communication System (PECS), an AAC system designed to minimize difficulties with communication skills experienced by individuals with Autism Spectrum Disorder | 30 Sessions ( 2 Months)
  The Picture Exchange Communication System (PECS) is an AAC system designed specifically to minimize difficulties with communication skills experienced by individuals with ASD. Presently, aided, picture-based AAC systems are used more frequently and successfully with individuals with ASD. PECS consists of six phases and begins by teaching an individual to give a single picture of a desired item or action to a "communicative partner" who immediately honors the exchange as a request. The system goes on to teach discrimination of pictures and how to put them together in sentences. In the more advanced phases, individuals are taught to use modifiers, answer questions and comment. The primary goal of PECS is to teach functional communication. It is a treatment choice for teaching speech to non-verbal children with autism but there is little empirical evidence available regarding the usefulness of picture exchange communication system in managing social and communication issues in autism.

CONTACTS AND LOCATIONS:
Overall Officials: Nameeka Shahid, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thiemann-Bourque K, Brady N, McGuff S, Stump K, Naylor A. Picture Exchange Communication System and Pals: A Peer-Mediated Augmentative and Alternative Communication Intervention for Minimally Verbal Preschoolers With Autism. J Speech Lang Hear Res. 2016 Oct 1;59(5):1133-1145. doi: 10.1044/2016_JSLHR-L-15-0313. PMID 27679841
- [Background] Lord C, Brugha TS, Charman T, Cusack J, Dumas G, Frazier T, Jones EJH, Jones RM, Pickles A, State MW, Taylor JL, Veenstra-VanderWeele J. Autism spectrum disorder. Nat Rev Dis Primers. 2020 Jan 16;6(1):5. doi: 10.1038/s41572-019-0138-4. PMID 31949163
- [Background] Ganz JB, Simpson RL. Effects on communicative requesting and speech development of the Picture Exchange Communication System in children with characteristics of autism. J Autism Dev Disord. 2004 Aug;34(4):395-409. doi: 10.1023/b:jadd.0000037416.59095.d7. PMID 15449515
- [Background] Mukherjee SB. Autism Spectrum Disorders - Diagnosis and Management. Indian J Pediatr. 2017 Apr;84(4):307-314. doi: 10.1007/s12098-016-2272-2. Epub 2017 Jan 19. PMID 28101829